CLINICAL TRIAL: NCT03216980
Title: Examining the Effect of Mental Health Disorders on Vascular Function and Exercise Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HM20009929
Record Dates: First submitted 2017-06-27; First posted 2017-07-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Mental Health Disorders
Keywords: cardiovascular disease; vascular function; PTSD; GAD
MeSH Terms: conditions — Cardiovascular Diseases; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PTSD/GAD Antioxidant (Experimental): Subjects will ingest an antioxidant cocktail containing 800 milligrams of alpha lipoic acid, 1 gram of vitamin C (ascorbic acid), and 400 milligrams of vitamin E (alpha tocopherol).
  Interventions: Dietary Supplement: PTSD/GAD Antioxidant; Dietary Supplement: PTSD/GAD Placebo
- PTSD/GAD Placebo (Placebo Comparator): Subjects will ingest placebo (microcrystalline cellulose) pills.
  Interventions: Dietary Supplement: PTSD/GAD Antioxidant; Dietary Supplement: PTSD/GAD Placebo
- Healthy Control Antioxidant (Experimental): Subjects will ingest an antioxidant cocktail containing 800 milligrams of alpha lipoic acid, 1 gram of vitamin C (ascorbic acid), and 400 milligrams of vitamin E (alpha tocopherol).
  Interventions: Dietary Supplement: Healthy Control Antioxidant; Dietary Supplement: Healthy Control Placebo
- Healthy Control Placebo (Placebo Comparator): Subjects will ingest placebo (microcrystalline cellulose) pills.
  Interventions: Dietary Supplement: Healthy Control Antioxidant; Dietary Supplement: Healthy Control Placebo

INTERVENTIONS:
Dietary Supplement: PTSD/GAD Antioxidant — Subjects will ingest an antioxidant cocktail containing 800 milligrams of alpha lipoic acid, 1 gram of vitamin C (ascorbic acid), and 400 milligrams of vitamin E (alpha tocopherol).
  Arms: PTSD/GAD Antioxidant; PTSD/GAD Placebo
Dietary Supplement: PTSD/GAD Placebo — Subjects will ingest placebo (microcrystalline cellulose) pills.
  Arms: PTSD/GAD Antioxidant; PTSD/GAD Placebo
Dietary Supplement: Healthy Control Antioxidant — Subjects will ingest an antioxidant cocktail containing 800 milligrams of alpha lipoic acid, 1 gram of vitamin C (ascorbic acid), and 400 milligrams of vitamin E (alpha tocopherol).
  Arms: Healthy Control Antioxidant; Healthy Control Placebo
Dietary Supplement: Healthy Control Placebo — Subjects will ingest placebo (microcrystalline cellulose) pills.
  Arms: Healthy Control Antioxidant; Healthy Control Placebo

SUMMARY:
Specific Aim #1: Examining the impact of mental health disorders (PTSD and GAD) on peripheral vascular function and sympathetic nervous system activity in young individuals.

Specific Aim #2: Examining the impact of mental health disorders (PTSD and GAD) on peripheral hemodynamics and metabolic byproducts during small muscle mass exercise in young individuals.

Specific Aim #3: Examining the impact of mental health disorders (PTSD and GAD) on exercise tolerance, peripheral hemodynamics and metabolic byproducts during large muscle mass exercise in young individuals.

DETAILED DESCRIPTION:
Mental health disorders are highly prevalent and underdiagnosed and can cause perturbations in cardiovascular and metabolic function leading to substantial individual burden (increased health care cost, loss of work productivity). Post-traumatic stress disorder (PTSD) and generalized anxiety disorder (GAD), two common mental health disorders, can cause increase cardiovascular disease risk due to chronic increases or fluctuations in heart rate, blood pressure, stress hormones, inflammation, and oxidative stress. Post-traumatic stress disorder (PTSD) is a disabling psychiatric condition characterized by a persistent maladaptive reaction resulting from exposure to severe psychological stress. It has been revealed that individuals with PTSD, in addition to adverse mental health symptoms, also possess higher prevalence rates for physical comorbidities such as hypertension, obesity, diabetes, and metabolic syndrome. Taken together, these PTSD-induced comorbidities result in a significant increase in the likelihood of developing cardiovascular disease (CVD) when compared to individuals without PTSD. Anxiety disorders, the most prevalent mental health issue in the United States, is associated an increased incidence of hypertension and heart disease. This increased cardiovascular disease (CVD) risk is thought to derive from an overactivation of the sympathetic nervous system that results in a predominately pro-oxidant, pro-inflammatory cardiovascular environment. Peripheral vascular dysfunction, or the inability of the blood vessels to adequately respond to specific stimuli, is a factor closely related to CVD. Therefore, this study will focus on a younger population with PTSD or GAD in an attempt to ascertain the presence of peripheral vascular dysfunction and the magnitude to which two potential primary contributors (autonomic dysfunction, oxidative stress) are involved in this dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy and free of overt cardiovascular, pulmonary, or metabolic disease
* for PTSD group, a score of ≥ 33 on PCL-5 checklist
* for GAD group, a score of ≥ 10 on the GAD-7 self-report scale

Exclusion Criteria:

* taking medications that could influence cardiovascular function
* limited English proficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Arm Vascular Function at Rest (Flow Mediated Dilation Test) and in Response to Exercise (Handgrip Exercise Test) | Before and Immediately After Intervention
  Change in Brachial Artery Dilation from Baseline Values
Leg Vascular Function (Passive Leg Movement Test) | Before and Immediately After Intervention
  Change in Leg Blood Flow Values from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Garten, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States